CLINICAL TRIAL: NCT05728177
Title: Effect of Inhalation Aromatherapy on Anxiety and Depressive Symptoms of Geriatric Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1112023
Record Dates: First submitted 2023-02-04; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Inhalation Aromatherapy
Keywords: Inhalation Aromathrapy, Anxiety, Depressive Symptoms, Parkinson's Disease
MeSH Terms: conditions — Anxiety Disorders; Depression; Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STUDY GROUP (Experimental): Patients' medical charts in the outpatient clinic were reviewed to identify those who meet the inclusion criteria. Patients who meet the predetermined inclusion criteria were recruited in the study using simple randomization technique using computer-generated sequence technique to pick up these patients. After simple sampling and dividing patients into two groups of study and control. Patients from the study and control groups were interviewed individually by the researcher to apply the study tools
  The program of intervention took four-weeks for each patient (total eight sessions- four outpatient sessions and four home-based sessions- two sessions per week- one outpatient and one home session/week). The outpatient sessions were done once per week during the patient visit to the outpatient clinic, as the patients visited the clinic 4 times/ month.
  Interventions: Combination Product: Inhalation Aromatherapy
- Control group (Active Comparator): Patients in this control group will be left without any intervention to undergo the usual outpatient routine care.
  Interventions: Combination Product: Inhalation Aromatherapy

INTERVENTIONS:
Combination Product: Inhalation Aromatherapy — Aromatherapy is safe, well prepared mixture used in the study that prepared by professor of pharmacology, faculty of pharmacy by mixing lavender essential oil and lavender hydrolate
  Patients' medical charts in the outpatient clinic were reviewed to identify those who meet the inclusion criteria. Patients who meet the predetermined inclusion criteria were recruited in the study using simple randomization technique using computer-generated sequence technique to pick up these patients. After simple sampling and dividing patients into two groups of study and control. Patients from the study and control groups were interviewed individually by the researcher to apply the study tools as a pretest. Aromatherapy intervention was carried out for patients in the study group while those in the control group were left without any intervention to undergo the usual outpatient routine care.

SUMMARY:
The present study aims to:

Investigate the effect of inhalation aromatherapy on anxiety and depressive symptoms of geriatric patients with Parkinson's disease.

Research Hypothesis:

Patients with Parkinson's disease who inhale aromatherapy will exhibit lower anxiety and depressive symptoms than those who didn't inhale it

DETAILED DESCRIPTION:
A sample of 60 randomly selected patients with patients Parkinson's disease was included in this study. The study subjects were divided equally into two groups; study (30 patients) and a control group (30 patients) matched as much as possible. Exclusion criteria included patients diagnosed for Parkinson's by a specialist, no use of any complementary alternative medicine methods (herbal medicines and other methods) in the past one week, no use of anxiolytics or antidepressants drugs, no history of respiratory problems as asthma, eczema and allergies to flowers and plants and no smell disorders. Patients who were not willing to participate, not able to provide written consent or not able to communicate coherently and relevantly or showed symptoms of allergy to lavender were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

patients diagnosed for Parkinson's by a specialist

Exclusion Criteria:

no use of any complementary alternative medicine methods (herbal medicines and other methods) in the past one week, no use of anxiolytics or antidepressants drugs, no history of respiratory problems as asthma, eczema and allergies to flowers and plants and no smell disorders. Patients who were not willing to participate, not able to provide written consent or not able to communicate coherently and relevantly or showed symptoms of allergy to lavender will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
The Beck Depression Inventory (BDI-II) | 2 weeks
  The scale was developed by (Beck, 1979; Beck, Steer, & Brown, 1996a; Beck, Ward, Mendelson, Mock, & Erbaugh, 1961). It is a standardized self-report rating inventory that measures attitudes and symptoms of depression in normal and populations with psychiatric disorders. The BDI-II contains 21 items across two Affective and Somatic subscales. Each item is measured on a 4-point Likert scale from 0 (symptom absent) to 3 (severe symptoms). In addition, items of sleep and appetite were assessed over seven options to determine their hypo or hyperactivity level. The minimum score is 0, and the maximum score is 63, while higher scores indicate greater severity of depressive symptoms. The total score of 0-13 is considered the minimal range of depressive symptoms; 14-19 is mild; 20-28 is moderate, and 29-63 is severe.

OTHER OUTCOMES:
Beck Anxiety Inventory (BAI) | 2 weeks
  The Beck Anxiety Inventory (BAI) was developed in 1988 and consists of 21 items with a Likert scale ranging from 0 to 3 and raw scores ranging from 0 to 63 (Beck, Epstein, Brown, & Steer, 1988). The questions used in this measure ask about common symptoms of anxiety that the subject has had during the past week (including the day you take it). The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The scores are classified as low anxiety (0-21), moderate anxiety (22-35) and potentially concerning levels of anxiety for score of 36 and above

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marsh L. Depression and Parkinson's disease: current knowledge. Curr Neurol Neurosci Rep. 2013 Dec;13(12):409. doi: 10.1007/s11910-013-0409-5. PMID 24190780
- [Result] Tang SK, Tse MY. Aromatherapy: does it help to relieve pain, depression, anxiety, and stress in community-dwelling older persons? Biomed Res Int. 2014;2014:430195. doi: 10.1155/2014/430195. Epub 2014 Jul 13. PMID 25114901